CLINICAL TRIAL: NCT04721457
Title: Mouth Rinses Efficacy on Salivary SARS-CoV-2 Viral Load: A Randomized Clinical Trial
Brief Title: The Efficacy of Pre-procedural Mouth Rinses on COVID-19 Saliva Viral Load
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, MANAR ALZAHRANI, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-02-J-002; 1384
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2; COVID-19; Mouthwashes; Viral Load; Polymerase Chain Reaction; Coronavirus; Covid19; Saliva
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Water; Povidone-Iodine; Mouthwashes; Hydrogen Peroxide; Cetylpyridinium; hydrated silica gel-based toothpaste; Sodium Hypochlorite

STUDY DESIGN:
Intervention Model Description: This randomizeda, single-center, randomized, double-blind, six-parallel-group, placebo-controlled trial compares the efficacy of four commercially available mouth rinses povidone-iodine (PVP-I), hydrogen peroxide (H2O2), cetylpyridinium chloride (CPC), sodium hypochlorite (NaOCl) on the salivary SARS-CoV-2 viral load at four-time points (baseline and 5-, 30-, and 60-min post rinsing) relative to two control groups (distilled water and no-rinse) in a cohort of positive COVID-19 patients.
Who Masked: Participant, Investigator
Masking Description: Allocated mouth rinses will be concealed in opaque sealed envelopes. Each envelope contains a 15 ml sterile amber test tube filled with the assigned mouth rinse, a 120 ml sterile empty specimen container for expectoration of the mouth rinse, and four identical empty 50 ml sterile test tubes for collecting saliva samples, each labeled with the allocated number and time point (T0, T1, T2, or T3), and a biohazard bag.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Distilled Water (Placebo Comparator): Vigorously rinse with 15 ml of the distilled water for 30 s (Water for Injections BP; Pharmaceutical Solutions Industry, Jeddah, SA)
  Interventions: Drug: Distilled Water
- Povidone Iodine (PVP-I) (Active Comparator): Vigorously rinse with 15 ml of the 1% povidone-iodine (PVP-I) (Betadine Mouthwash/Gargle; Avrio Health LP, Stamford, CT, USA) for 30 s
  Interventions: Drug: 1% Povidone Iodine (PVP-I)
- Hydrogen Peroxide (H2O2) (Active Comparator): Vigorously rinse with 15 ml of the 1.5% hydrogen peroxide (H2O2) (Peroxyl; Colgate-Palmolive, Guildford, UK) for 30 s
  Interventions: Drug: 1.5% Hydrogen Peroxide (H2O2)
- Cetylpyridinium Chloride (CPC) (Active Comparator): Vigorously rinse with 15 ml of the 0.075% cetylpyridinium chloride (CPC) (Colgate Total; Colgate-Palmolive, Guildford, UK) for 30 s
  Interventions: Drug: 0.075% Cetylpyridinium Chloride (CPC)
- Sodium Hypochlorite (Active Comparator): Vigorously rinse with 15 ml of the 80 ppm sodium hypochlorite (NaOCl) (Clinisept Dental Mouthwash; Clinical Health Technologies, Hinckley, Leicestershire, UK) for 30 s
  Interventions: Drug: 0.1% Sodium Hypochlorite
- No rinse group (Placebo Comparator): There is no mouth rinse in this group. Patients will collect the saliva at all 4-time points without gargling with the mouth rinse.
  Interventions: Other: No rinse group

INTERVENTIONS:
Drug: Distilled Water — Control group
  Other Names: water (Water for Injections BP; Pharmaceutical Solutions Industry, Jeddah, SA)
  Arms: Distilled Water
Drug: 1% Povidone Iodine (PVP-I) — Over-the-counter antiseptic mouth rinse
  Other Names: Betadine Mouthwash/Gargle; Avrio Health LP, Stamford, CT, USA
  Arms: Povidone Iodine (PVP-I)
Drug: 1.5% Hydrogen Peroxide (H2O2) — Over-the-counter antiseptic mouth rinse
  Other Names: Peroxyl; Colgate-Palmolive, Guildford, UK
  Arms: Hydrogen Peroxide (H2O2)
Drug: 0.075% Cetylpyridinium Chloride (CPC) — Over-the-counter antiseptic mouth rinse
  Other Names: Colgate Total; Colgate-Palmolive, Guildford, UK
  Arms: Cetylpyridinium Chloride (CPC)
Drug: 0.1% Sodium Hypochlorite — Over-the-counter antiseptic mouth rinse
  Other Names: Clinisept Dental Mouthwash; Clinical Health Technologies, Hinckley, Leicestershire, UK
  Arms: Sodium Hypochlorite
Other: No rinse group — second control group
  Arms: No rinse group

SUMMARY:
Preoperative antiseptic mouth rinses have been widely used as a standard protocol before routine dental treatment reduces oral microorganism counts. During dental procedures, aerosolized microorganisms contaminate the dental environment and nearby surfaces and remain suspended for 4 hours. Thus, the reduction in the number of aerosolized microorganisms by pre-procedural rinsing may reduce cross-contamination between dentists, office personnel, and patients. Recent reviews have advocated the use of preoperative rinsing to control and reduce the risk of SARS-CoV-2 transmission. However, no clinical studies have been done yet to support the effectiveness of any pre-procedural oral rinses against SARS-CoV-2. The proposed study will mitigate the spread of COVID-19 disease in dental healthcare facilities and ensure the patients' good health and healthcare workers. The purpose of this clinical trial is to compare the efficacy of four commercially available mouth rinses povidone-iodine (PVP-I), hydrogen peroxide (H2O2), cetylpyridinium chloride (CPC), sodium hypochlorite (NaOCl) on the salivary SARS-CoV-2 viral load at four-time points (baseline and 5-, 30-, and 60-min post rinsing) relative to two control groups (distilled water and no-rinse) in a cohort of positive COVID-19 patients.

DETAILED DESCRIPTION:
Saliva specimens will be collected from COVID-19-positive patients presenting to TETAMMAN clinics from January to March 2021. The total number of participants in this study will be 90 participants, with 15 per group (6 groups), and 4 saliva specimens from each patient in each group. A total of four mouth rinses and two control groups (distilled water and no-rinse). The studied mouth rinses were: 1% povidone-iodine (PVP-I) (Betadine Mouthwash/Gargle; Avrio Health LP, Stamford, CT, USA), 1.5% hydrogen peroxide (H2O2) (Peroxyl; Colgate-Palmolive, Guildford, UK), 0.075% cetylpyridinium chloride (CPC) (Colgate Total; Colgate-Palmolive, Guildford, UK), 80 ppm sodium hypochlorite (NaOCl) (Clinisept Dental Mouthwash; Clinical Health Technologies, Hinckley, Leicestershire, UK). Confirmed positive cases of COVID-19 will be recruited randomly at each TETAMMAN clinic based on inclusion and exclusion criteria to satisfy the total of 90 patients. Each participant will be introduced briefly to the study aims and then asked to sign a consent form. Demographic data and medical history will then be collected for each participant. The participants will be blinded to all mouth rinses, which will be labeled with identification codes, and presented in similar packages. Unstimulated saliva will be collected using the passive drool technique. Four saliva samples for each patient will be collected. The first saliva sample will be considered as a baseline sample that represents the baseline viral load. Then patients will be instructed to gargle the assigned mouth rinse gently, for 15 seconds. After that, the participants will spit the mouthwashes into a disposable plastic cup. After that, different salivary samples will be collected at 5 minutes, 30 minutes, and then 60 minutes. Thus, a total of four saliva samples will be gathered from each patient. The viral load will be measured by quantitative reverse transcription PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years or older presented to TETAMMAN clinics, Jeddah, Saudi Arabia.
2. COVID-19-positive patients confirmed by RT-PCR and within two days of oral or nasopharyngeal swabs
3. Asymptomatic or within seven days of the onset of symptoms.
4. Has the ability to rinse and expectorate.

Exclusion Criteria:

1. Participants who established antiviral, corticosteroid, antimicrobial, or immunosuppressive medications.
2. Known allergy to one of the constituents of the mouth rinse
3. Thyroid disease or on current radioactive iodine treatment
4. Pregnant or breastfeeding women
5. Lithium therapy
6. History of radiotherapy or chemotherapy
7. Use of mouthwash before presented to TETAMMAN clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in the salivary viral load within each mouth rinse groups and controls | Baseline (T0) vs 5 minutes (T1), baseline (T0) vs 30 minutes (T2), and baseline (T0) vs 60 minutes T3)
  change in the salivary viral load overtime within each group will be measured by quantitative reverse transcription PCR (RT-qPCR) and expressed as copies/ml
Compare salivary viral load between mouth rinse groups and controls at baseline | Compare Baseline (T0)
  Difference in Salivary viral load baseline value between the groups
Compare salivary viral load between mouth rinse groups and controls at 5 minutes post rinsing | 5 minutes post rinsing (T1)
  Difference in Salivary viral load baseline value between the groups
Compare salivary viral load between mouth rinse groups and controls at 30 minutes post rinsing | 30 minutes post rinsing (T2)
  Difference in Salivary viral load baseline value between the groups
Compare salivary viral load between mouth rinse groups and controls at 60 minutes post rinsing | 60 minutes post rinsing (T3)
  Difference in Salivary viral load baseline value between the groups

CONTACTS AND LOCATIONS:
Overall Officials: MANAR M ALZAHRANI, MSD, FRCD(C), Principal Investigator — King Abdulaziz University
Locations (1):
- Alhamra TETAMMAN clinic (PHC), Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Result] Ge ZY, Yang LM, Xia JJ, Fu XH, Zhang YZ. Possible aerosol transmission of COVID-19 and special precautions in dentistry. J Zhejiang Univ Sci B. 2020 May;21(5):361-368. doi: 10.1631/jzus.B2010010. Epub 2020 Mar 16. PMID 32425001
- [Result] Vergara-Buenaventura A, Castro-Ruiz C. Use of mouthwashes against COVID-19 in dentistry. Br J Oral Maxillofac Surg. 2020 Oct;58(8):924-927. doi: 10.1016/j.bjoms.2020.08.016. Epub 2020 Aug 15. PMID 32859459
- [Result] O'Donnell VB, Thomas D, Stanton R, Maillard JY, Murphy RC, Jones SA, Humphreys I, Wakelam MJO, Fegan C, Wise MP, Bosch A, Sattar SA. Potential Role of Oral Rinses Targeting the Viral Lipid Envelope in SARS-CoV-2 Infection. Function (Oxf). 2020;1(1):zqaa002. doi: 10.1093/function/zqaa002. Epub 2020 Jun 5. PMID 33215159
- [Result] Carrouel F, Conte MP, Fisher J, Goncalves LS, Dussart C, Llodra JC, Bourgeois D. COVID-19: A Recommendation to Examine the Effect of Mouthrinses with beta-Cyclodextrin Combined with Citrox in Preventing Infection and Progression. J Clin Med. 2020 Apr 15;9(4):1126. doi: 10.3390/jcm9041126. PMID 32326426
- [Result] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Result] Bruch MK. Toxicity and safety of topical sodium hypochlorite. Contrib Nephrol. 2007;154:24-38. doi: 10.1159/000096812. PMID 17099299
- [Result] De Nardo R, Chiappe V, Gomez M, Romanelli H, Slots J. Effects of 0.05% sodium hypochlorite oral rinse on supragingival biofilm and gingival inflammation. Int Dent J. 2012 Aug;62(4):208-12. doi: 10.1111/j.1875-595X.2011.00111.x. Epub 2012 May 11. PMID 23017003
- [Result] Seo HW, Seo JP, Cho Y, Ko E, Kim YJ, Jung G. Cetylpyridinium chloride interaction with the hepatitis B virus core protein inhibits capsid assembly. Virus Res. 2019 Apr 2;263:102-111. doi: 10.1016/j.virusres.2019.01.004. Epub 2019 Jan 9. PMID 30639191
- [Result] Feres M, Figueiredo LC, Faveri M, Stewart B, de Vizio W. The effectiveness of a preprocedural mouthrinse containing cetylpyridinium chloride in reducing bacteria in the dental office. J Am Dent Assoc. 2010 Apr;141(4):415-22. doi: 10.14219/jada.archive.2010.0193. PMID 20354090
- [Result] Marui VC, Souto MLS, Rovai ES, Romito GA, Chambrone L, Pannuti CM. Efficacy of preprocedural mouthrinses in the reduction of microorganisms in aerosol: A systematic review. J Am Dent Assoc. 2019 Dec;150(12):1015-1026.e1. doi: 10.1016/j.adaj.2019.06.024. PMID 31761015
- [Result] Pitten FA, Kramer A. Efficacy of cetylpyridinium chloride used as oropharyngeal antiseptic. Arzneimittelforschung. 2001;51(7):588-95. doi: 10.1055/s-0031-1300084. PMID 11505791
- [Result] Osso D, Kanani N. Antiseptic mouth rinses: an update on comparative effectiveness, risks and recommendations. J Dent Hyg. 2013 Feb;87(1):10-8. Epub 2013 Feb 5. PMID 23433693
- [Result] Caruso AA, Del Prete A, Lazzarino AI. Hydrogen peroxide and viral infections: A literature review with research hypothesis definition in relation to the current covid-19 pandemic. Med Hypotheses. 2020 Nov;144:109910. doi: 10.1016/j.mehy.2020.109910. Epub 2020 Jun 1. PMID 32505069
- [Result] Walsh LJ. Safety issues relating to the use of hydrogen peroxide in dentistry. Aust Dent J. 2000 Dec;45(4):257-69; quiz 289. doi: 10.1111/j.1834-7819.2000.tb00261.x. PMID 11225528
- [Result] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Result] Kariwa H, Fujii N, Takashima I. Inactivation of SARS coronavirus by means of povidone-iodine, physical conditions and chemical reagents. Dermatology. 2006;212 Suppl 1(Suppl 1):119-23. doi: 10.1159/000089211. PMID 16490989